CLINICAL TRIAL: NCT05045963
Title: Evaluating the Impact of Aminoglycosides in Hypotensive Septic Oncology Patients
Brief Title: Impact of Aminoglycosides in Hypotensive Septic Oncology Patients
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-0999; NCI-2021-01105 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0999 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-03-01; First posted 2021-09-16 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm; Septicemia
MeSH Terms: conditions — Hematologic Neoplasms; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational (medical record review): Patients' medical charts are reviewed retrospectively.
  Interventions: Other: Electronic Health Record Review

INTERVENTIONS:
Other: Electronic Health Record Review — Medical record reviewed

SUMMARY:
This study evaluates the impact of aminoglycosides in hypotensive septic oncologic patients. In the oncologic patient population, sepsis is a major health concern due to high mortality rates and healthcare costs. Prior research shows aminoglycosides antibiotics are frequently used to treat sepsis, but their clinical impact in hypotensive oncology patients upon the progression of sepsis is not known.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the impact of beta-lactam (BL) + aminoglycoside (AG) combination therapy in hypotensive septic oncology patients.

OUTLINE:

Patients' medical charts are reviewed retrospectively.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age >= 18 years) with a diagnosis of sepsis during the index hospital admission identified by International classification of diseases (ICD)-10 codes (as specified below) receiving BL antibiotics within 6 hours prior to or following the onset of hypotension
* To be included in the AG group, patients must have received at least 1 dose of intravenous (IV) tobramycin or amikacin in addition to the BL therapy within the above time period

Exclusion Criteria:

* Age < 18 years
* Receipt of IV AG outside of the above time frame in the AG group or receipt of IV AG within 48 hours prior to or following the onset of hypotension in the BL backbone group
* Pregnancy
* Patients not receiving therapy with BL antibiotics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Oncology patients with sepsis and hypotension treated at The University of Texas MD Anderson Cancer Center from January 1, 2019 to December 31, 2019
Sampling Method: Non-Probability Sample
Enrollment: 319 (Estimated)
Dates: Start 2021-01-04 (Actual); Primary Completion 2025-09-21 (Estimated); Study Completion 2025-09-21 (Estimated)

PRIMARY OUTCOMES:
Time to resolution of hypotension | Within 7 days from hypotension onset
  Defined as a mean arterial pressure > 65 mmHg not requiring vasopressors and sustained for >= 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey J Bruno, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center — http://www.mdanderson.org